CLINICAL TRIAL: NCT04420585
Title: Desmopressin as a Therapy for Nocturnal Enuresis in Pediatric Patients With Sickle Cell Disease
Brief Title: Desmopressin for Bedwetting in Children With SCD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not able to meet recruitment after 9 years of trying to enroll patients on different versions of the protocol and changing recruitment strategies.
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11268
Record Dates: First submitted 2020-05-21; First posted 2020-06-09 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Nocturnal Enuresis; Anemia, Sickle Cell
MeSH Terms: conditions — Nocturnal Enuresis; Anemia, Sickle Cell | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Desmopressin 0.2mg tablets, dose titrated to effect
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Two desmopressin 0.2 mg tablets at bedtime for 14 days and monitoring if <50 % improvement
  Other Names: DDAVP

SUMMARY:
This study assesses if using the medication desmopressin will decrease nightime bedwetting in children with sickle cell disease.

DETAILED DESCRIPTION:
Night time bedwetting is a common complication of sickle cell disease, and affects up to 30 % of children. Desmopressin is an oral medication that increases water reabsorption in the kidneys. Studies have shown that it is effective in decreasing bedwetting episodes in children without sickle cell disease. Chronic sickling episodes causing damage to the kidneys could cause permanent damage and may make this treatment ineffective in sickle cell disease. This trial will inform pediatric sickle cell doctors if desmopressin is an appropriate treatment for bed wetting in the investigators patients.

This study expanded upon a previously terminated study which had separately registered (NCT02636387, ID: 2014-3768).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Hemoglobin SS, SC, SB0thal or SB+thal
2. Patients with at least two episodes of primary nocturnal enuresis per week or four episodes over the two weeks prior to enrollment.
3. Patients with secondary enuresis who have been evaluated and cleared by a pediatric urologist as not having other etiologies of enuresis (e.g. overactive detrusor activity, a genitourinary anatomic abnormality)

Exclusion Criteria:

1. Patients with developmental delay or neurologic dysfunction secondary to stroke.
2. Patients with hypertension or underlying renal disease.
3. Patients with genitourinary anatomic abnormalities. Any prior renal ultrasound showing normal genitourinary anatomy is sufficient to clear a patient for the study.
4. Patients with daytime urinary incontinence
5. Patients with glucosuria on urinalysis.
6. Patients with secondary nocturnal enuresis who have not been evaluated by a pediatric urologist to rule out other etiologies of enuresis.
7. Patients who are pregnant.
8. Patients receiving another medicine for nocturnal enuresis (e.g. imipramine).

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Morrone, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Children's Hospital at Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neveus T, von Gontard A, Hoebeke P, Hjalmas K, Bauer S, Bower W, Jorgensen TM, Rittig S, Walle JV, Yeung CK, Djurhuus JC. The standardization of terminology of lower urinary tract function in children and adolescents: report from the Standardisation Committee of the International Children's Continence Society. J Urol. 2006 Jul;176(1):314-24. doi: 10.1016/S0022-5347(06)00305-3. PMID 16753432
- [Background] Barakat LP, Smith-Whitley K, Schulman S, Rosenberg D, Puri R, Ohene-Frempong K. Nocturnal enuresis in pediatric sickle cell disease. J Dev Behav Pediatr. 2001 Oct;22(5):300-5. doi: 10.1097/00004703-200110000-00004. PMID 11718233
- [Background] Readett DR, Morris JS, Serjeant GR. Nocturnal enuresis in sickle cell haemoglobinopathies. Arch Dis Child. 1990 Mar;65(3):290-3. doi: 10.1136/adc.65.3.290. PMID 2334206
- [Background] Field JJ, Austin PF, An P, Yan Y, DeBaun MR. Enuresis is a common and persistent problem among children and young adults with sickle cell anemia. Urology. 2008 Jul;72(1):81-4. doi: 10.1016/j.urology.2008.02.006. Epub 2008 Apr 2. PMID 18384865
- [Background] Naitoh Y, Kawauchi A, Soh J, Kamoi K, Miki T. Health related quality of life for monosymptomatic enuretic children and their mothers. J Urol. 2012 Nov;188(5):1910-4. doi: 10.1016/j.juro.2012.07.012. Epub 2012 Sep 19. PMID 22999692
- [Background] Glazener CM, Evans JH. Desmopressin for nocturnal enuresis in children. Cochrane Database Syst Rev. 2002;(3):CD002112. doi: 10.1002/14651858.CD002112. PMID 12137645
- [Background] Becker AM. Sickle cell nephropathy: challenging the conventional wisdom. Pediatr Nephrol. 2011 Dec;26(12):2099-109. doi: 10.1007/s00467-010-1736-2. Epub 2011 Jan 4. PMID 21203778
- [Background] Statius van Eps LW, Schouten H, Haar Romeny-Wachter CC, La Porte-Wijsman LW. The relation between age and renal concentrating capacity in sickle cell disease and hemoglobin C disease. Clin Chim Acta. 1970 Mar;27(3):501-11. doi: 10.1016/0009-8981(70)90305-0. No abstract available. PMID 5435231
- [Background] Figueroa TE, Benaim E, Griggs ST, Hvizdala EV. Enuresis in sickle cell disease. J Urol. 1995 Jun;153(6):1987-9. PMID 7752379
- [Background] Robson WL, Leung AK, Norgaard JP. The comparative safety of oral versus intranasal desmopressin for the treatment of children with nocturnal enuresis. J Urol. 2007 Jul;178(1):24-30. doi: 10.1016/j.juro.2007.03.015. Epub 2007 May 11. PMID 17574054

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Desmopressin 0.2mg tablets, dose titrated to effect
  NOTE: While an option, doses were not titrated for any of the participants in this study prior to study termination.
  Desmopressin: Two desmopressin 0.2 mg tablets at bedtime for 14 days and monitoring if <50 % improvement
Period: Overall Study
Arm/Group | Treatment Group
Started | 8
Completed | 5
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Never initiated medication | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Genotype of Sickle Cell Disease [Count of Participants; unit: Participants] — The number of participants with Sickle Cell Anemia (Hb SS) vs Sickle Hemoglobin-C (Hb SC) was determined.
  Participants
    Sickle Cell Anemia (Hb SS) | 6
    Sickle Hemoglobin-C Disease (Hb SC) | 2
Number of Bedwetting Days Based on Disease Type [Mean (Standard Deviation); unit: days] — Participants were asked to recall the number of days during which a bedwetting episode was experienced over the prior 14 days. Mean number of days was reported by disease type. Population: 6 participants had Sickle Cell Anemia (Hb SS) and two participants had Sickle Hemoglobin-C (Hb SC)
  days
    Sickle Cell Anemia (Hb SS): number analyzed (Participants) | 6
    Sickle Cell Anemia (Hb SS) | 10.5 (4.0)
    Sickle Hemoglobin-C Disease (Hb SC): number analyzed (Participants) | 2
    Sickle Hemoglobin-C Disease (Hb SC) | 8.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bedwetting Episodes
Description: Change in the percentage of nights with bedwetting episodes assessed at baseline based on participant recall over the previous 14 nights, as well as at ~1 month (30 nights) based on completion of a study (enuresis) diary. This is used to assess whether the use of desmopressin in patients with sickle cell disease and nocturnal enuresis will decrease the number of nighttime episodes of enuresis by 50% after initiating DDAVP at 0.4 mg nightly dose (with dose escalation as clinically appropriate). A negative value indicates a decrease in bedwetting episodes.
Time Frame: Baseline and ~1 month
Measure: Mean (Standard Deviation); unit: percentage of nights
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
percentage of nights | -41 (26.2)

2. Secondary Outcome: Impact of Bedwetting on Day to Day Activities
Description: To determine if patients with sickle cell disease and nocturnal enuresis receiving desmopressin will have an improved quality of life compared to their baseline. This will be measured using the PedsQL Measurement Model which measures health related quality of life in children with acute and chronic health conditions, like sickle cell. The scales focuses on areas such as activities, feelings, and school performance.
Time Frame: Baseline and 4 weeks
Population: Data was not collected for the Impact of Bedwetting on day-to-day activities.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Nighttime Awakenings
Description: Change in the percentage of nights with awakenings over the previous 14 nights was assessed by summarizing and comparing baseline and 1 month nighttime awakening data. The percentage of nights with nighttime awakenings was evaluated at baseline based on recall and at 1 month (30 nights) based on completion of a study diary. This was used to determine whether the use of desmopressin in patients with sickle cell disease and nocturnal enuresis changes the rates of nighttime awakenings to urinate (nocturia), defined as episodes of nighttime awakening to void in children ≥5 years of age, compared to prior to initiating treatment with DDAVP. A positive value indicates an increase in nighttime awakenings
Time Frame: Baseline and ~1 month
Measure: Mean (Standard Deviation); unit: percentage of nights
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
percentage of nights | 16.8 (25.3)

4. Secondary Outcome: Change in Daytime Fatigue
Description: Change in daytime fatigue will be assessed to determine if patients with sickle cell disease and nocturnal enuresis receiving desmopressin will have less daytime fatigue compared to their baseline data. The PROMIS Pediatric Fatigue Short Form (Version 2.0) will be used to compare levels of fatigue from baseline and ~1 month (30 nights) on the study medication. The PROMIS Fatigue scale, which utilizes a 7-day recall period, is a 10-item questionnaire consisting of 5 responses ranging from 1-5 with one indicative of "Never" and five indicative of "almost always" resulting in a raw scoring range of 10-50. Negative PROMIS change scores are associated with decreased levels of fatigue.
Time Frame: Baseline and ~1 month
Population: 1 month fatigue data was not able to collected from one participant who did not complete the 1 month PROMIS Fatigue questionnaire. Accordingly, change results were not available.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
score on a scale | -6.0 [-18 to 6]

ADVERSE EVENTS:
Time Frame: 4 weeks after initiation of medication
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=8)
Dizziness (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT04420585/Prot_SAP_000.pdf